CLINICAL TRIAL: NCT06494410
Title: Comparison of the Effect of High Versus Low Fraction of Inspired Oxygen During Alveolar Recruitment on Absorption Atelectasis in Laparoscopic Bariatric Surgery Patients With Atelectasis
Brief Title: Effect of High Versus Low Fraction of Inspired Oxygen During Alveolar Recruitment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Abdallah Adel Saber
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2023-02

CONDITIONS: Bariatric Surgery Candidate; Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Fraction of Inspired Oxygen(Group A) (Active Comparator): About 40 patients received FiO2 1.0 during recruitment maneuvers
  Interventions: Procedure: High versus Low Fraction of Inspired Oxygen
- Low Fraction of Inspired Oxygen(Group B) (Active Comparator): About 40 patients received FiO2 0.4 during recruitment maneuvers
  Interventions: Procedure: High versus Low Fraction of Inspired Oxygen

INTERVENTIONS:
Procedure: High versus Low Fraction of Inspired Oxygen — to compare the effect of high oxygen fraction (FiO2 1.0) vs. low oxygen fraction (FiO2 0.4) on clinical outcome on intraoperative and postoperative atelectasis and PPC. We will asses the impact of FiO2, especially during RM, on atelectasis development, using modified LUSS in obese patients with atelectasis undergoing laparoscopic bariatric surgery.

SUMMARY:
Intraoperative absorption atelectasis is associated with decreased lung compliance, impaired oxygenation, increased pulmonary vascular resistance, and lung injury.

The alveolar recruitment maneuver (RM) with positive-end expiratory pressure (PEEP) has been advocated as efficient for absorption atelectasis treatment.

During general anesthesia, absorption atelectasis reportedly occurs in most patients especially during laparoscopic surgery, the increased abdominal pressure of capnoperitoneum may shift the diaphragm cranially and decrease respiratory compliance

DETAILED DESCRIPTION:
The incidence of obesity (defined by a body mass index (BMI) > 30 kg/m2) is increasing worldwide. In selected individuals, bariatric surgery may offer means of achieving long-term weight loss, improved health, and healthcare cost reduction. Physiological changes that occur because of obesity and general anesthesia predispose to respiratory complications following bariatric surgery.

Obesity affects many respiratory functions, including, among others, a reduction in functional residual capacity, an increase in airway resistance, and a high level of ventilation-perfusion mismatch. The combination of obesity and postoperative respiratory muscle dysfunction could promote respiratory failure.

Absorption atelectasis occurs in most patients, typically due to absorption of gas, compression of the lung tissue, and impairment of surfactant function. Additionally, during laparoscopic surgery, the increased abdominal pressure of capnoperitoneum may shift the diaphragm cranially and decrease respiratory compliance.

Compression of basal lung regions due to a stiffened diaphragm would accelerate the formation of absorption atelectasis that was already initiated during anesthesia induction.

Such deterioration is associated with pulmonary densities revealed by computed tomography. In addition to physiologic impairment, atelectasis could contribute to perioperative lung injury and PPC.

The RM with PEEP has been advocated as efficient for atelectasis treatment. Reports on the impact of FiO2 during RM on atelectasis development are rare, and have not limited FiO2 to the RM per se.

While RM with high FiO2 can improve oxygenation rapidly, there is a greater possibility of absorption atelectasis occurring.

Diagnostic ultrasonography is the only clinical imaging technology in use that does not depend on electromagnetic radiation. Lung ultrasonography can be considered an attractive complementary diagnostic tool and one of the most promising techniques (Daabis et al., 2014). Therefore, Lung ultrasonography is a safe and cheap tool used during the perioperative period and to detect intraoperative respiratory complications resulting from absorption atelectasis.

The modified Lung Ultrasound Score (LUSS) system involves examination of all intercostal spaces: each hemi-thorax is divided into six regions: 2 anterior, 2 lateral and 2 posterior with four longitudinal lines and one axial line [figure 1 (B, C)]. Each region score shows sufficient sensitivity to detect loss of aeration during laparoscopic surgery. The degree of de-aeration rated from 0 to 3 (zero for no atelectasis and 3 for complete atelectasis ) defining substantial atelectasis as a score of 2 or 3 assigned to any region

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 - 60 years old.
* Both genders.
* Preoperative Physical Status: ASA II, III Patients.
* BMI above 40 Kg/m2.
* Patients undergoing laparoscopic bariatric surgeries: laparoscopic mini gastric bypass, Roux-en-Y gastric bypass and revision bariatric surgery (redo bariatric surgery) with the presence of atelectasis confirmed radiologically by Chest X-ray (CXR) and CT Chest

Exclusion Criteria:

* Refusal of the intervention or participation in the study.
* Patient under age of 18 years old or above 60 years old.
* Preoperative Physical Status: ASA I, IV.
* Psychiatric illness.
* Known cases of chronic pulmonary disease e.g. COPD and bronchial asthma.
* Known cases of cardiac diseases.
* Previous lung surgery.
* Lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Modified Lung Ultrasound Score (LUSS) | from 0 hours to 6 hours after the procedure
  1. Modified LUSS at surgery completion compared to baseline preoperative modified LUSS, reflecting any aeration loss during general anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Madiha Metwaly Zidan, Professor, Study Chair — Department of Anesthesia and I.C.U. faculty of Medicine,Ain Shams university, Egypt; Ahmed Ali Fawaz, Professor, Study Director — Department of Anesthesia and I.C.U. faculty of Medicine,Ain Shams university, Egypt
Locations (1):
- Ain Shams University Hospitals, Cairo, Abbasia, Egypt